CLINICAL TRIAL: NCT01849159
Title: Clinical Study of the Efficacy and Safety of the Application of Allogeneic Mesenchymal (Stromal) Cells of Bone Marrow, Cultured Under the Hypoxia in the Treatment of Patients With Severe Pulmonary Emphysema
Status: Withdrawn | Phase: Phase 1 / Phase 2 | Type: Interventional
Sponsor: Federal Research Clinical Center of Federal Medical & Biological Agency, Russia (Other Government)
Responsible Party: Principal Investigator, Alexander Averyanov, Deputy of Director General of FRCC, Federal Research Clinical Center of Federal Medical & Biological Agency, Russia
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: MSC-HYP-01; FMBA-FRCC-MSC-01 (Other: Federal Medical&Biological Agency)
Record Dates: First submitted 2013-04-24; First posted 2013-05-08 (Estimated); Last update posted 2018-01-09 (Actual); Status verified 2018-01

CONDITIONS: Pulmonary Emphysema
Keywords: Mesenchymal stem cells; Hypoxia; Emphysema
MeSH Terms: conditions — Pulmonary Emphysema; Hypoxia; Emphysema

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- MSC group (Active Comparator): Intravenous infusion of MSC suspension, pre-conditioned under 1% oxygen, in the amount of 200 mln. cells per 400 mL of sodium chloride physiological solution. Infusions will be performed every 2 months for 1 year
  Interventions: Biological: Mesenchymal stem cells
- Control Group (Placebo Comparator): 400 mL of 0.9% NaCl solution. Infusions will be performed every 2 months for 1 year
  Interventions: Other: Reference therapy: 400 mL of 0.9% NaCl solution

INTERVENTIONS:
Biological: Mesenchymal stem cells — Intravenous infusion of MSC suspension, pre-conditioned under 1% oxygen, in the amount of 200 mln. cells per 400 mL of sodium chloride physiological solution
  Arms: MSC group
Other: Reference therapy: 400 mL of 0.9% NaCl solution
  Arms: Control Group

SUMMARY:
Actively developing stem cells (SCs) transplantation techniques cause natural interest to the problem of regeneration in the lungs. Numerous experimental studies proved the benefits of different types of SCs in experimental models of pulmonary emphysema (PE).

G. Zhen et al. have shown that the transplantation of mesenchymal stem cells (MSCs) to rats with papain-induced emphysema leads to their migration into the lungs, differentiation into type 2 alveolocytes, and inhibition of apoptosis and prevention PE.

K. Schweitzer et al. have proved the activity of inflammation in the airways, alveolocytes and endothelial cells apoptosis decreased after adipose SCs intravenous administration to mice with emphysema caused by chronic exposure to tobacco smoke or VEGF receptors blockade. The study of E.P. Ingenito et al. found that endobronchial installed MSCs engraft into the alveolar wall and peribronchial interstitium and release integrins, extracellular matrix components (collagen IV, laminin and fibrillin), platelet-derived growth factor receptor and transforming growth factor β2.

Our study also found reliable deterrent effect of allogeneic bone marrow MSCs on the development of elastase-induced emphysema in rats at different terms of transplantation.

After the success of pilot studies have started clinical trials. Currently, the website http://www. ClinicalTrials.gov reported three studies evaluating the efficacy and safety of MSC transplantation in patients with COPD and emphysema. Two of them have already been completed and the results of the first pilot project published.

Authors on the example of 4 patients showed a complete absence of adverse effects, improved quality of life and stability of functional parameters at 12 months after starting treatment One of the problems of MSC transplantation in patients with respiratory failure is an accelerated apoptosis of transplanted cells under the influence of proinflammatory cytokines and oxidative stress. Since it is proved that preconditioning MSCs under hypoxia increases their survival in hypoxic conditions, increases the expression of growth factors and antiinflammatory cytokines, we suppose that MSCs grown in hypoxic medium may have a significant positive effect on the disease.

ELIGIBILITY:
Inclusion Criteria:

* HRCT-confirmed diagnosis of lung emphysema by two independent radiologists
* post-bronchodilator FEV1/FVC ratio < 0.7
* post-bronchodilator FEV1 % predicted value ≥ 20% and < 50%
* age 35 and 75 years of, of either sex, and of any race
* current or ex-smoker, with a cigarette smoking history ≥ 10 pack-years

Exclusion Criteria:

* • asthma or other clinically relevant lung disease other than COPD (e.g. restrictive lung diseases, sarcoidosis, tuberculosis, idiopathic pulmonary fibrosis, or lung cancer)

  * α1-Antitrypsin deficiency
  * Presence of bullae (more than 10 cm in the diameter)
  * active infection within 4 weeks of screening
  * significant exacerbation of COPD or has required mechanical ventilation within 4 weeks of screening
  * clinically relevant uncontrolled medical condition not associated with COPD
  * documented history of uncontrolled heart failure
  * pulmonary hypertension due to left heart condition
  * Subject has evidence of active malignancy, or prior history of active malignancy
  * Subject has a life expectancy of < 6 months

Ages: 35 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 0 (Actual)
Dates: Start 2014-03; Primary Completion 2016-12 (Estimated); Study Completion 2017-06 (Estimated)

PRIMARY OUTCOMES:
Safety compared with placebo | 1 year
  Mortality (Baseline and 2 years after procedure) Adverse effects and reactions to the treatment(Baseline and 2 years after procedure).
  Vital signs (pulse rate, systolic and diastolic arterial blood pressure) (Baseline and 2 years after procedure)

SECONDARY OUTCOMES:
Change from baseline in the lung tissue density measured by CT-densitometry at6, 12, 24 months | 2 years
DLCO change from baseline at 6, 12, 24 months | 2 years
Change from baseline in the functional parameters (FEV1, TLC, RV, FEV1/FVC) at 6,12,18,24 months | 2 years
Dynamics of the physical capacity (by the 6-min test results) | 2 years
Dynamics of the blood gas composition (PaO2, PaCO2) | 2 years
Dynamics of serum level IL-6, TNF-α, Leptin | 2 years
Quality of life indices by the questionnaire (SF-36) | 2 years
Number and frequency of exacerbations | 2 years
Body mass index | 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Alexander V Averyanov, MD, PhD, Principal Investigator — Federal Research Clinical Center of Federal Medical and Biological Agency
Locations (1):
- Federal Research Clinical Center of Federal Medical and Biological Agency of Russia, Moscow, Moscow Oblast, Russia